CLINICAL TRIAL: NCT04767646
Title: Evaluation of the Relationship Between the Duration of the Evolution of the Complex Regional Pain Syndrome Type 1 (CRPS 1) and Effectiveness of the Continuous Peripheral Nerve Block (CPNB) Associated With an Intensive Rehabilitation Program
Acronym: BLOCALGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00084-35
Record Dates: First submitted 2021-02-05; First posted 2021-02-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: CRPS (Complex Regional Pain Syndrome) Type I
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-BNP with intensive rehabilitation program (Experimental)
  Interventions: Procedure: Intensive rehabilitation program with CPNB

INTERVENTIONS:
Procedure: Intensive rehabilitation program with CPNB — The patient will have an intensive rehabilitation program (two 30-minute kinesitherapy sessions every day and 30-minute occupational therapy sessions 5 days a week) with the CPNB.
  The patient will have follow-up consultation at 1 month, 3 month, 6 month and 1 year after the beggining of the intensive rehabilitation program

SUMMARY:
The study evaluates the relationship between the duration of evolution of SDRC1 and the efficacy of continuous peripheral nerve block (c-PNB) associated with an intensive rehabilitation program to improve the therapeutic strategy of SDRC1.

The main hypothesis of this study is that if c-PNB is proposed earlier, the recovery, measured with a scale achievement of objectives, will be better.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* Diagnosis of CRPS type 1 according to BUDAPEST criteria to the upper or lower limb
* Affiliated to a social security scheme (beneficiary or entitled person)
* Patients justifying the installation of a Continuous Peripheral Nerve Block (CPNB) including pain rebellious to physical and medicinal treatments, the presence of fixed dystonia, or kinesiphobia or who are no longer progressing in the rehabilitation algorithm and requiring the need for a specialised technical platform.

Exclusion Criteria:

* CRPS Type 2
* Contra-indication to the analgesics used (bupivacaine, ropivacaine, levobupivacaine)
* Severe psychiatric decompensation
* Under legal protection measures
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The composite score (the summation of the 3 Goal Attainment Scaling (GAS) scores) | 1 year
  The improvement of the composite score following BNPc combined with intensive rehabilitation.

SECONDARY OUTCOMES:
Pain assessment | 1 year
  EVA (Visual Analogue Scale, VAS) for all the patients at each visit This is a measure of pain intensity on a scale of 0 (no pain) to 10 (very severe pain).
  We will assess the percentage of pain relief with the EVA scale, before and after the PCNB.
Anxiety assessment | 1 year
  Hospital Anxiety and Depression (HAD) scale for all the patients at each visit There will be 2 scores One to assess anxiety : from 0 to 21 and one to assess depression : from 0 to 21 Higher scores mean a worse outcome.
Arthrometry assessment | 1 year
  For an upper limb block :
  Passive and active arthrometry (angular measurements for shoulder, elbow and wrist)
  For a block of the lower limb :
  Passive and active arthrometry (angular measurements for hip, knee and ankle)
hand joint assessment | 1 year
  For an upper limb block :
  Kapandji Index at each visit (between 0 to 10)
gripping force assessment | 1 year
  For an upper limb block, gripping force will be evaluated with a Jamar and Pinch dynamometer at each visit after BNPc
activity assessment | 1 year
  For an upper limb block, the activity limitation will be evaluated by leroux's scapular index (LSI) with a global score out of 100 at each visit after BNPc
manual dexterity test | 1 year
  For an upper limb block, the dexterity will be evaluated by a Box and Block Test at each visit after BNPc
Assessment of activity limitation for a block of the upper limb | 1 year
  DASH scale at each visit
Assessment of activity limitation for a block of the lower limb | 1 year
  WOMAC score at each visit
Assessment of functional capacity | 1 year
  TDM6 at each visit (number of metres travelled by the patient during 6 minutes)
Assessment of the restriction of participation in social life | 1 year
  Return to work
Evaluation of the effective dose | During the CPNB
  - Recording of effective doses (continuous and bolus)
Evaluation of the tolerance of CPNB | During the CPNB
  - Incident reporting

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pôle Saint Hélier, Rennes, Brittany Region, France